CLINICAL TRIAL: NCT02555592
Title: Treatment Strategy of Surgical Resection With Sequential Adjuvant Chemotherapy and Radiotherapy for Patients With Stage IIIA Non-small Cell Lung Cancer and N2 Disease Only in the Subaortic or Paraaortic Level, or Both
Brief Title: Strategy of Surgical Resection With Adjuvant Therapy for IIIA NSCLC and N2 Disease Only in Subaortic or Paraaortic Level
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Jung Seop Eom, Clinical assistant professor, Pusan National University Hospital
Other Study IDs: 56 study
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Lung Cancer; Cancer of Lymph Node; Effects of Chemotherapy; Surgery
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Primary surgical resection with sequential adjuvant therapy — First, surgery resection of the affected lung with mediastinal lymph node dissection, including sub- and para-aortic lymph node, will be performed. If malignant tumor involvement only in the sub- or para-aortic lymph nodes is identified, adjuvant chemotherapy will be initiated within 8 weeks after surgery. After completion of adjuvant chemotherapy, post-operative radiotherapy will be initiated within 2~4 weeks after adjuvant chemotherapy.

SUMMARY:
The purpose of this study is to identify the treatment outcomes of surgical resection with sequential adjuvant chemotherapy and radiotherapy in patients with stage IIIA non-small cell lung cancer and N2 disease at only the sub- or para-aortic level.

DETAILED DESCRIPTION:
Stage IIIA non-small cell lung cancer (NSCLC) is a very heterogeneous disease and current treatment guidelines recommend concurrent chemoradiation therapy or combined neoadjuvant chemotherapy, surgical resection, and sequential adjuvant therapy. When incidental N2 disease is found despite thorough preoperative staging, adjuvant platinum-based chemotherapy with or without adjuvant radiotherapy is recommended.

Although guidelines suggest preoperative mediastinal staging with endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA), this method does not allow approach of the sub- or para-aortic lymph nodes. Therefore, patients with suspected stage IIIA NSCLC and N2 disease only at the sub- or para-aortic level should undergo several processes if combined neoadjuvant chemotherapy and surgical resection is planned. First, video-assisted thoracoscopic surgery (VATS) should be performed to verify whether the sub- or para-aortic lymph nodes are involved. If a frozen-section biopsy reveals no malignant tumor involvement in the sub- and para-aortic lymph nodes, the affected lung can be resected. If there is sub- or para-aortic lymph node involvement, further neoadjuvant chemotherapy is required before surgical resection and adjuvant therapy.

Studies have shown that stage IIIA NSCLC with only sub- or para-aortic lymph node involvement has better outcomes than other stage IIIA NSCLC. Moreover, the five-year survival of patients with stage IIIA NSCLC with only sub- or para-aortic lymph node involvement is similar to that with stage II NSCLC. However, those studies were retrospective with relatively small sample sizes. Therefore, we evaluated the outcomes of combined surgical resection with adjuvant chemotherapy and radiotherapy in patients with stage IIIA NSCLC and N2 disease at only the sub- or para-aortic level.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IIIA non-small cell lung cancer and suspicious of N2 disease only in the subaortic or paraaortic level, or both on chest CT or PET scan

Exclusion Criteria:

* Patients whose subaortic or paraaortic lymph nodes were revealed as negative by mediastinal lymph node dissection
* Patients whose mediastinal lymph nodes other than subaortic or paraaortic level were confirmed as malignant node by mediastinal lymph node dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage IIIA non-small cell lung cancer and N2 disease only in the subaortic or paraaortic level, or both
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2015-10; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Three-year disease free survival | Three year

SECONDARY OUTCOMES:
Three-year survival rate | Three year
Five-year survival rate | Five year
Recurrence rate | Five year

CONTACTS AND LOCATIONS:
Overall Officials: Jung Seop Eom, Master, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Busan, Busan, South Korea

REFERENCES:
- [Background] Silvestri GA, Gonzalez AV, Jantz MA, Margolis ML, Gould MK, Tanoue LT, Harris LJ, Detterbeck FC. Methods for staging non-small cell lung cancer: Diagnosis and management of lung cancer, 3rd ed: American College of Chest Physicians evidence-based clinical practice guidelines. Chest. 2013 May;143(5 Suppl):e211S-e250S. doi: 10.1378/chest.12-2355. PMID 23649440
- [Background] Vansteenkiste J, De Ruysscher D, Eberhardt WE, Lim E, Senan S, Felip E, Peters S; ESMO Guidelines Working Group. Early and locally advanced non-small-cell lung cancer (NSCLC): ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2013 Oct;24 Suppl 6:vi89-98. doi: 10.1093/annonc/mdt241. Epub 2013 Jul 16. No abstract available. PMID 23860613
- [Background] De Leyn P, Dooms C, Kuzdzal J, Lardinois D, Passlick B, Rami-Porta R, Turna A, Van Schil P, Venuta F, Waller D, Weder W, Zielinski M. Revised ESTS guidelines for preoperative mediastinal lymph node staging for non-small-cell lung cancer. Eur J Cardiothorac Surg. 2014 May;45(5):787-98. doi: 10.1093/ejcts/ezu028. Epub 2014 Feb 26. PMID 24578407
- [Background] Cerfolio RJ, Bryant AS, Eloubeidi MA. Accessing the aortopulmonary window (#5) and the paraaortic (#6) lymph nodes in patients with non-small cell lung cancer. Ann Thorac Surg. 2007 Sep;84(3):940-5. doi: 10.1016/j.athoracsur.2007.04.078. PMID 17720403
- [Background] Miller DL, McManus KG, Allen MS, Ilstrup DM, Deschamps C, Trastek VF, Daly RC, Pairolero PC. Results of surgical resection in patients with N2 non-small cell lung cancer. Ann Thorac Surg. 1994 May;57(5):1095-100; discussion 1100-1. doi: 10.1016/0003-4975(94)91335-8. PMID 8179370
- [Background] Nakanishi R, Osaki T, Nakanishi K, Yoshino I, Yoshimatsu T, Watanabe H, Nakata H, Yasumoto K. Treatment strategy for patients with surgically discovered N2 stage IIIA non-small cell lung cancer. Ann Thorac Surg. 1997 Aug;64(2):342-8. doi: 10.1016/S0003-4975(97)00535-3. PMID 9262572
- [Background] Okada M, Tsubota N, Yoshimura M, Miyamoto Y, Matsuoka H. Prognosis of completely resected pN2 non-small cell lung carcinomas: What is the significant node that affects survival? J Thorac Cardiovasc Surg. 1999 Aug;118(2):270-5. doi: 10.1016/S0022-5223(99)70217-5. PMID 10425000
- [Background] Keller SM, Vangel MG, Wagner H, Schiller JH, Herskovic A, Komaki R, Marks RS, Perry MC, Livingston RB, Johnson DH; Eastern Cooperative Oncology Group. Prolonged survival in patients with resected non-small cell lung cancer and single-level N2 disease. J Thorac Cardiovasc Surg. 2004 Jul;128(1):130-7. doi: 10.1016/j.jtcvs.2003.11.061. PMID 15224032